CLINICAL TRIAL: NCT00956449
Title: A Phase II, Single Center, Uncontrolled, Open-Label Study to Evaluate Safety and Immunogenicity of a Surface Antigen, Inactivated Influenza Vaccine [Ph.Eur], Formulation 2009/2010, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of Influenza Vaccine (Surface Antigen, Inactivated) [Ph.Eur], Formulation 2009-2010, When Administered to Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Novartis, Novartis Vaccines
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V78_07S; 2009-011004-33
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Influenza; Seasonal Influenza
Keywords: flu; influenza; seasonal influenza; influenza vaccine antigen; immunogenicity; safety; tolerability; antibody response; intra muscular; elderly; non-elderly
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Seasonal Influenza Vaccine

INTERVENTIONS:
Biological: Seasonal Influenza Vaccine — 1 dose of Influenza Vaccine Surface Antigen, Inactivated

SUMMARY:
The purpose of this study is to evaluate the antibody response to each of the three influenza vaccine strains included in the licensed seasonal flu vaccine, as measured by hemagglutination inhibition (HI) at 21 days post immunization in non-elderly and elderly subjects in compliance with the requirements of the current European Union (EU) recommendations for the evaluation of the immunogenicity for a new formulation of a licensed flu vaccine (CPMP/BWP/214/96).

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for enrollment into this study are male and female adults who are:

  * ≥ 18 years of age, mentally competent, willing and able to give informed consent prior to study entry;
  * able to comply with all study requirements;
  * in good health as determined by:

    1. medical history,
    2. physical examination,
    3. clinical judgment of the investigator.

Exclusion Criteria:

* Subjects are not to be enrolled into the study if at least one of the following criteria is fulfilled:

  * They have any serious chronic or acute disease (in the judgment of the investigator) including but not limited to:

    1. Cancer, except for localized skin cancer
    2. Advanced congestive heart failure
    3. Chronic obstructive pulmonary disease (COPD)
    4. Autoimmune disease (including rheumatoid arthritis)
    5. Acute or progressive hepatic disease
    6. Acute or progressive renal disease
    7. Severe neurological or psychiatric disorder
    8. Severe Asthma
  * History of any anaphylactic reaction and/or serious allergic reaction following a vaccination, a proven hypersensitivity to any component of the study vaccine (e.g., to eggs, chicken protein, chicken feathers, influenza viral protein neomycin or polymyxin).
  * Known or suspected (or have a high risk of developing) impairment/alteration of immune function (excluding that normally associated with advanced age) resulting for example from:

    1. receipt of immunosuppressive therapy (any parental or oral cortical steroid or cancer chemotherapy/radiotherapy) within the past 60 days and for the full length of the study;
    2. Receipt of immunostimulants,
    3. Receipt of parenteral immunoglobulin preparation, blood products, and/or plasma derivatives within the past 3 months and for the full length of the study,
    4. Suspected or known HIV infection or HIV-related disease.
  * Known or suspected history of drug or alcohol abuse.
  * They have a bleeding diathesis or conditions associated with prolonged bleeding time that in the investigator's opinion would interfere with the safety of the subject;
  * Women who are pregnant or woman of childbearing potential unwilling to practice acceptable contraception for the duration of the study (21 days). Females who are pregnant or nursing (breastfeeding) mothers or females of childbearing age who do not plan to use acceptable birth control measures, for the duration of the study. Adequate contraception is defined as hormonal (oral, injection, transdermal patch, implant, cervical ring), barrier (condom or diaphragm), intrauterine device (IUD) or monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject's study entry.
  * Influenza vaccination or laboratory confirmed influenza within the last 6 months and more than one influenza vaccination within the past 12 months
  * Within the past 4 weeks they have received: another vaccine or any investigational agent.
  * Any acute or chronic infection requiring systemic antibiotic treatment or antiviral therapy within the last 7 days.
  * They have experienced fever (i.e., axillary temperature ≥ 38°C) within the last 3 days
  * Simultaneous participation in another clinical study.
  * Any condition, which, in the opinion of the investigator, might prevent the subject from participation or interfere with the evaluation of the study objectives.
  * Severely obese with Body Mass Index (BMI) > 35
  * Site personnel involved in evaluation of safety and their immediate relatives are excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity and tolerability of the Flu vaccines is being measured | 2 - 21 days

SECONDARY OUTCOMES:
To evaluate safety of a single IM (intramuscular) dose of the subunit vaccine of Influenza Vaccine Surface Antigen, Inactivated of Influenza Vaccine | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (1):
- The Health Centre, Suffolk, United Kingdom